CLINICAL TRIAL: NCT00908609
Title: 3-D Simultaneous Ultrasound and NIR Imaging for Breast Cancer Detection
Brief Title: Optical Tomography With Ultrasound Guidance
Status: Completed | Type: Observational
Sponsor: UConn Health (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Donaghue Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Quing Zhu, Professor, UConn Health
Other Study IDs: 02-064S-2; R01EB002136 (NIH)
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Diagnosis; Optical Imaging; Ultrasound Imaging; Monitoring Neoadjuvant Chemotherapy Response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients who undergo routine ultrasound guided biopsy will be studied by optical imaging technique.
- 2: Patients who have advanced breast cancers and are under neoadjuvant chemotherapy treatment will be studied by optical technique.

SUMMARY:
The investigators propose to validate the utility of their novel hybrid imaging technique for accurate diagnosis of breast lesions, and for assessing chemotherapy response of cancer treatment and predicting treatment efficacy. The investigators' unique hybrid technique is implemented by simultaneously deploying near infrared (NIR) optical sensors and a commercial ultrasound (US) transducer mounted on a hand-held probe, and utilizing co-registered lesion structure information provided by ultrasound to improve the optical tomography.

As a result, the optical tomography assisted with US has overcome problems associated with intense light scattering and has provided reliable tumor angiogenesis distributions. Initial results with a small group of patients who underwent biopsy have shown that early stage invasive cancers present two-fold greater total hemoglobin concentration on average than fibroadenomas and other benign lesions. Initial results of advanced cancers have shown that the angiogenesis distribution is highly distorted and heterogeneous, and the distorted distributions correlate with histological microvessel density counts and can be used to assess chemotherapy response.

The objective of this study is to validate the investigators' initial results that NIR light guided by ultrasound can improve breast cancer diagnosis and monitor chemotherapy response.

DETAILED DESCRIPTION:
Specific objectives of the study are:

Objective 1: Validate the sensitivity, specificity, positive predictive value and negative predictive value of optical tomography/US for distinguishing benign and early stage malignant breast tumors. Approximately 300 patients who will undergo ultrasound-guided biopsy are being recruited to this study from the University of Connecticut Health Center and Hartford Hospital. The total hemoglobin concentration and blood oxygen saturation will be the measured indices and the biopsy results will be used as the 'gold' standard.

Objective 2: Perform pilot studies of optical tomography/US to assess chemotherapy response and evaluate treatment efficacy. Patients diagnosed with locally advanced breast cancers (size greater than 3 cm) who will undergo chemotherapy will be enrolled to this study. Approximately, 20 to 30 patients are being recruited to the study from the University of Connecticut Health Center and Hartford Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing ultrasound guided biopsy or breast cancer patients undergoing neoadjuvant thermotherapy treatment

Exclusion Criteria:

* Women under 18 years old.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Women undergo ultrasound guided biopsy
  2. Breast cancer patients undergo neoadjuvant thermotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2007-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The deoxygenated/oxygenated hemoglobin and total hemoglobin concentration are the measured imaging parameters and biopsy results will be used as the 'gold' standard to compare imaging findings. | 4 more years

CONTACTS AND LOCATIONS:
Overall Officials: Quing Zhu, Ph.D, Principal Investigator — University of Connecticut
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut

REFERENCES:
- [Result] Zhu Q, Hegde PU, Ricci A Jr, Kane M, Cronin EB, Ardeshirpour Y, Xu C, Aguirre A, Kurtzman SH, Deckers PJ, Tannenbaum SH. Early-stage invasive breast cancers: potential role of optical tomography with US localization in assisting diagnosis. Radiology. 2010 Aug;256(2):367-78. doi: 10.1148/radiol.10091237. Epub 2010 Jun 22. PMID 20571122
- [Result] Xu Y, Zhu Q. Imaging heterogeneous absorption distribution of advanced breast cancer by optical tomography. J Biomed Opt. 2010 Nov-Dec;15(6):066007. doi: 10.1117/1.3505015. PMID 21198181
- [Result] Xu C, Zhu Q. Light shadowing effect of large breast lesions imaged by optical tomography in reflection geometry. J Biomed Opt. 2010 May-Jun;15(3):036003. doi: 10.1117/1.3431086. PMID 20615005
- [Result] Ardeshirpour Y, Huang M, Zhu Q. Effect of the chest wall on breast lesion reconstruction. J Biomed Opt. 2009 Jul-Aug;14(4):044005. doi: 10.1117/1.3160548. PMID 19725717
- [Result] Xu C, Yuan B, Zhu Q. Optimal probe design for breast imaging using near-infrared diffused light. J Biomed Opt. 2008 Jul-Aug;13(4):044002. doi: 10.1117/1.2966703. PMID 19021330
- [Result] Zhu Q, Tannenbaum S, Hegde P, Kane M, Xu C, Kurtzman SH. Noninvasive monitoring of breast cancer during neoadjuvant chemotherapy using optical tomography with ultrasound localization. Neoplasia. 2008 Oct;10(10):1028-40. doi: 10.1593/neo.08602. PMID 18813360
- [Result] Zhu Q, Wang L, Tannenbaum S, Ricci A Jr, DeFusco P, Hegde P. Pathologic response prediction to neoadjuvant chemotherapy utilizing pretreatment near-infrared imaging parameters and tumor pathologic criteria. Breast Cancer Res. 2014 Oct 28;16(5):456. doi: 10.1186/s13058-014-0456-0. PMID 25349073
- [Result] Tavakoli B, Zhu Q. Two-step reconstruction method using global optimization and conjugate gradient for ultrasound-guided diffuse optical tomography. J Biomed Opt. 2013 Jan;18(1):16006. doi: 10.1117/1.JBO.18.1.016006. PMID 23296038
- [Result] Zhu Q, DeFusco PA, Ricci A Jr, Cronin EB, Hegde PU, Kane M, Tavakoli B, Xu Y, Hart J, Tannenbaum SH. Breast cancer: assessing response to neoadjuvant chemotherapy by using US-guided near-infrared tomography. Radiology. 2013 Feb;266(2):433-42. doi: 10.1148/radiol.12112415. Epub 2012 Dec 21. PMID 23264349